CLINICAL TRIAL: NCT04261140
Title: Clinical Evaluation of Four Aesthetic Restorations in Non-carious Cervical Lesions: a Randomised Controlled Split-mouth Clinical Trial
Brief Title: Clinical Evaluation of Four Aesthetic Restorations in Non-carious Cervical Lesions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: required license
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gul Yildiz Telatar, Principal Investigator, Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/19
Record Dates: First submitted 2020-02-04; First posted 2020-02-07 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Noncarious Cervical Lesions
Keywords: High-viscosity glass ionomer; bulkfill composite; flowable composite; nanohybrid composite; cervical lesion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High-viscosity glass ionomer (Experimental)
  Interventions: Other: EQUIA Forte Fil
- flowable composite (Experimental)
  Interventions: Other: NexComp Flow
- bulkfill composite (Experimental)
  Interventions: Other: 3M Espe Bulk-fill
- nanohybrid composite (Experimental)
  Interventions: Other: Clearfil Majesty Esthetic

INTERVENTIONS:
Other: EQUIA Forte Fil — Apply cavity conditioner (20% polyacrylic acid) 10 s on enamel and dentine, rinse Mix 10 s and apply bulk-fill Apply EQUIA coat and light cure for 20 s
  unit
  Arms: High-viscosity glass ionomer
Other: Clearfil Majesty Esthetic — Apply in 2-mm increment, light cure for 20 s
  Arms: nanohybrid composite
Other: NexComp Flow — Apply in 2-mm increment light cure for 20 s
  Arms: flowable composite
Other: 3M Espe Bulk-fill — Apply in single increment up to 4 mm; light curing for 20 s
  Arms: bulkfill composite

SUMMARY:
To compare the clinical performance of high-viscosity glass ionomer, flowable composite, bulkfill composite and nanohybrid composite restorations in non-carious cervical lesions (NCCLs).

DETAILED DESCRIPTION:
One hundred fourty NCCLs were randomised into four groups according to a split-mouth design. Clinical evaluations will be performed after 1 week, 3 months, 6 months, using FDI (World Dental Federation) criteria.

ELIGIBILITY:
Inclusion Criteria:

* had at least four non-carious symmetrical cervical lesions,
* had permanent dentition and were older than 20 years old,
* had cervical margins in dentin

Exclusion Criteria:

* periodontal disease
* pregnant or breastfeeding
* being under orthodontic therapy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
evaluation of restoration on cervical lesions | 6 months
  According to FDI criteria (aesthetic, biological and fuctional) score 1, clinically very good; score 2, clinically good; score 3, clinically sufficient; score 4, clinically unsatisfactory; score 5, clinically poor. Scores 1-3 show clinically acceptable restoration, while scores 4 and 5 indicate failure

CONTACTS AND LOCATIONS:
Overall Officials: Gül Yıldız Telatar, Dr, Principal Investigator — Recep Tayyip Erdogan University Dentistry Faculty
Locations (1):
- Recep Tayyip Erdogan University Dentistry Faculty, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be available within 1 years of study completion